CLINICAL TRIAL: NCT03902860
Title: Recording Sympathetic Nerve Activity From the Skin During Stellate, Thoracic, and Lumbar Sympathetic Ganglia Block : a Pilot Study
Brief Title: Measurement of the Skin Sympathetic Nerve Activity During Stellate, Thoracic, and Lumbar Sympathetic Ganglia Block
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor of Anesthesiology and Pain Medicine, Seoul National University Hospital
Other Study IDs: SGB SKNA pilot
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain Requiring Stellate, Thoracic, and Lumbar Sympathetic Ganglia Blockade

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sympathetic nerve activity can be measured transcutaneously in awake patients by computer-based filtering of raw signal obtained via skin leads attached on the chest and the right arm. Electrocardiogram can be removed by applying a high-pass filter setting of 150 Hz. Electromyogram can be filtered by applying a high-pass filter setting of 500 Hz or a band-pass filter setting of 500-1000 Hz.

Currently, the therapeutic effect of stellate, thoracic, and lumbar sympathetic ganglia block (SGB, TSGB, and LSGB, respectively) in patients with chronic pain is generally evaluated by using thermogram/thermography (change in temperature of the upper or lower extremeties) or questionnaire-based scoring.

However, it is not known whether the skin sympathetic nerve activity (SKNA) can be measured in patients undergoing SGB/TSGB/LSGB and used as an alternative tool for assessing the therapeutic effect of SGB/TSGB/LSGB.

Therefore, we planned this pilot study to observe whether the SKNA can be obtained in patients undergoing SGB/TSGB/LSGB and whether it is well correlated to thermogram or questionnaire-based scoring. If the SKNA is observed and decreases after SGB/TSGB/LSGB, it will be presented in milivolt (uV) and compared to that of pre-block values.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient patients undergoing stellate, thoracic, and lumbar sympathetic block for chronic pain disease

Exclusion Criteria:

* patients denial
* peripheral vascular disease in the head and the upper extremities.
* prior thoracic sympathectomy/sympathicotomy
* prior resection or ablation (chemically or mechanically) of stellate, thoracic, and lumbar sympathetic
* coagulapathy
* infectious disease
* allergy to local anesthetics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing stellate, thoracic, or lumbar sympathetic block for control of chronic neuropathic pain
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
The skin sympathetic nerve activity presented as uV obtained via skin leads. | From the beginning of stellate, thoracic, or lumbar sympathetic block procedure and the next outpatient visiting 4 weeks (an average) after the procedure.
  A few studies reported that skin sympathetic nerve activity (SKNA) signal could be potentially observed by applying a high-pass filter of 500 Hz or a band-pass filter of 500~1000 Hz to electric signal from skin leads attached on the skin of the chest in awake volunteers. However, it is not known if it would be also possible to observe the SKNA signal in patients undergoing stellate, thoracic, and lumbar sympathetic block. Also, there is no established, objective tool for quantitative or qualitative assessment of the effect of stellate, thoracic, and lumbar sympathetic block.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul National University Hospital, Seoul, South Korea